CLINICAL TRIAL: NCT03677869
Title: Single-Arm Study Assessing the Effects of Pneumatic Vitreolysis on Macular Hole
Brief Title: Effects of Pneumatic Vitreolysis on Macular Hole
Acronym: Protocol AH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DRCR.net Protocol AH; U10EY014231 (NIH)
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Results first posted 2021-06-29 (Actual); Last update posted 2022-09-19 (Actual); Status verified 2022-09

CONDITIONS: Vitreomacular Traction (VMT); Full-thickness Macular Holes (MH)
Keywords: Pneumatic Vitreolysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Pneumatic vitreolysis (PVL) (Experimental): Pneumatic vitreolysis is an in-office intraocular injection of an expansile gas (C3F8) to induce release of vitreomacular traction.
  Interventions: Device: Intraocular gas (C3F8)

INTERVENTIONS:
Device: Intraocular gas (C3F8) — Intraocular gas (C3F8) injection

SUMMARY:
Eyes with vitreomacular traction (VMT) and full-thickness macular holes (MH) will be enrolled into a non-randomized cohort treated with pneumatic vitreolysis (PVL) to determine the proportion with VMT release and MH closure and to assess factors associated with success.

DETAILED DESCRIPTION:
The objective of this trial is to obtain estimates of the proportion of eyes with MH closure of the inner retinal layers for eyes with VMT and full-thickness MHs treated with PVL. Understanding the rates of VMT release and MH closures in eyes with full-thickness MH treated with PVL is of interest. Surgery would result in nearly 100% hole closure and VMT release, making vitrectomy a poor control group choice. Spontaneous resolution of MH is highly unlikely, making an observation arm unnecessary. Therefore, these eyes will be enrolled into a non-randomized cohort treated with PVL to assess the outcomes of treatment.

ELIGIBILITY:
Participant-Level Criteria Inclusion

To be eligible, the following inclusion criteria must be met:

1. Age ≥ 18 years

   • Participants < 18 years old are not being included because the condition is so rare in this age group that the diagnosis may be questionable.
2. At least one eye meets the study eye criteria
3. Able and willing to provide informed consent
4. Able and willing to avoid high altitude travel, including airline travel, until gas resolution (approximately 6 to 8 weeks)
5. For phakic patients, able and willing to avoid supine position until gas resolution (approximately 6 to 8 weeks)
6. Able and willing to position face down for at least 50% of the time for at least 4 days post-injection (to facilitate macular hole closure)
7. Able and willing to wear wristband that informs any medical personnel that the patient has a gas bubble in the eye Exclusion

A potential participant is not eligible if any of the following exclusion criteria are present:

8. A condition that, in the opinion of the investigator, would preclude participation in the study (e.g., unstable medical status that might preclude completion of follow up) 9. Participation in an investigational trial within 30 days of enrollment that involves treatment with any drug or device that has not received regulatory approval for the indication being studied at the time of study entry

* Note: study participants should not receive another investigational drug or device while participating in the study 10. Known contraindication to any component of the treatment 11. Known allergy to any drug used in the procedure prep (including povidone iodine) 12. Potential participant is expecting to move out of the area of the clinical center to an area not covered by another clinical center during the 6 months following enrollment 13. Anticipated surgery requiring anesthesia within the 6 months following enrollment
* Participants cannot receive nitrous oxide until gas resolution 13. For women of child-bearing potential: pregnant at the time of enrollment
* Women who are potential study participants should be questioned about the potential for pregnancy. Investigator judgement may be used to determine when a pregnancy test is needed

Study Eye Criteria The participant must have at least one eye meeting all of the inclusion criteria and none of the exclusion criteria listed below.

A participant can have only one study eye. If both eyes are eligible at the time of enrollment, the study eye will be selected by the investigator and participant before injection.

The eligibility criteria for a study eye are as follows:

Inclusion

1. Full-thickness macular hole that is ≤ 250 microns at the narrowest point, confirmed by central reading center
2. Vitreomacular adhesion on OCT that is no larger than 3000 microns with visible separation of the vitreous on either side as seen on horizontal and vertical scans , confirmed by central reading center

   • Presence of epiretinal membrane is neither a requirement nor exclusion
3. Visual acuity letter score of at least 19 (approximate Snellen equivalent 20/400 or better) and at most 83 (20/25 or worse) Exclusion
4. Other ocular condition that might affect visual acuity during the course of the study or require intraocular treatment (e.g., retinal vein occlusion, substantial age-related macular degeneration, or macular edema induced by a condition other than VMT)

   * If diabetic retinopathy is present, severity level must be microaneurysms only or better (≤ diabetic retinopathy severity level 20).
   * Presence of drusen is acceptable; however, eyes with geographic atrophy or neovascular age-related macular degeneration involving the macula are excluded.
5. High level of myopia (spherical equivalent of -8.00 diopters or more myopic if phakic, or retinal abnormalities consistent with pathologic myopia if phakic or pseudophakic)
6. History of prior gas injection, ocriplasmin injection, or intraocular injection for any reason
7. History of prior vitrectomy
8. History of uncontrolled glaucoma

   • Intraocular pressure must be < 30 mmHg, with no more than one topical glaucoma medication, and no documented glaucomatous field loss for the eye to be eligible
9. History of major ocular surgery (including cataract extraction, scleral buckle, any intraocular surgery, etc.) within prior 4 months or major ocular surgery anticipated within the next 6 months following enrollment
10. History of YAG capsulotomy performed within 4 months prior to enrollment
11. Aphakia or anterior chamber intraocular lens
12. Exam evidence of severe external ocular infection, including conjunctivitis, chalazion, or substantial blepharitis
13. Uveitis
14. Retinal history or pathology that might predispose an eye to an increased risk of retinal detachment from the procedure

    • Untreated retinal tears, not retinal holes, are an exclusion. It is up to the investigator to determine whether extent of lattice degeneration or other pathology might increase the risk of retinal detachment
15. Any contraindication to paracentesis (e.g., history of narrow angle glaucoma)
16. Lenticular or zonular instability

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2018-11-14 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-07-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Calvin E Mein, MD, Study Chair — Retinal Consultants of San Antonio
Locations (45):
- United States (45):
  - Retinal Diagnostic Center, Campbell, California
  - Atlantis Eye Care, Huntington Beach, California
  - Northern California Retina Vitreous Associates, Mountain View, California
  - East Bay Retina Consultants, Inc., Oakland, California
  - Southern California Desert Retina Consultants, MC, Palm Desert, California
  - National Ophthalmic Research Institute, Fort Myers, Florida
  - University of Florida College of Med., Dept of Ophthalmology, Jacksonville Hlth Sci Ctr, Jacksonville, Florida
  - Florida Retina Consultants, Lakeland, Florida
  - Florida Retina Institute, Orlando, Florida
  - Southeast Eye Institute, PA dba Eye Associates of Pinellas, Pinellas Park, Florida
  - Retina Associates of Sarasota, Sarasota, Florida
  - Sarasota Retina Institute, Sarasota, Florida
  - Southeast Retina Center, PC, Augusta, Georgia
  - Thomas Eye Group, Sandy Springs, Georgia
  - Gailey Eye Clinic, Bloomington, Illinois
  - University of Illinois at Chicago Medical Center, Chicago, Illinois
  - Illinois Retina Associates, SC, Oak Park, Illinois
  - Carle Foundation Hospital, Urbana, Illinois
  - Raj K. Maturi, MD, PC, Indianapolis, Indiana
  - Wolfe Eye Clinic, West Des Moines, Iowa
  - Mid-America Retina Consultants, P.A., Overland Park, Kansas
  - Paducah Retinal Center, Paducah, Kentucky
  - Eye Associates of Northeast Louisiana dba Haik Humble Eye Center, West Monroe, Louisiana
  - Elman Retina Group, BA, Baltimore, Maryland
  - Valley Eye Physicians and Surgeons, Ayer, Massachusetts
  - Joslin Diabetes Center, Boston, Massachusetts
  - Vitreo-Retinal Associates, PC, Worcester, Massachusetts
  - Retina Specialists of Michigan, Grand Rapids, Michigan
  - Mayo Clinic Department of Ophthalmology, Rochester, Minnesota
  - The Retina Institute, St Louis, Missouri
  - MaculaCare, New York, New York
  - Retina-Vitreous Surgeons of Central New York, PC, Syracuse, New York
  - Western Carolina Clinical Research, LLC, Asheville, North Carolina
  - Charlotte Eye, Ear, Nose, and Throat Assoc., PA, Charlotte, North Carolina
  - Retina Associates of Cleveland, Inc., Beachwood, Ohio
  - Retina Vitreous Center, Edmond, Oklahoma
  - Oregon Retina, LLP, Eugene, Oregon
  - Retina Northwest, PC, Portland, Oregon
  - Southeastern Retina Associates, Chattanooga, Tennessee
  - Southeastern Retina Associates, PC, Knoxville, Tennessee
  - Austin Retina Associates, Austin, Texas
  - Retina Research Center, Austin, Texas
  - Medical Center Ophthalmology Associates, San Antonio, Texas
  - Retinal Consultants of San Antonio, San Antonio, Texas
  - Spokane Eye Clinic, Spokane, Washington

RESULTS

PARTICIPANT FLOW:
Recruitment Details: One eye that did not have full-thickness macular hole was enrolled, received PVL, and completed the 24-week visit but is not included in any analyses or subsequent levels in the participant flow
Period: Overall Study
Arm/Group | Pneumatic Vitreolysis (PVL)
Started | 35
Completed | 34
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Pneumatic Vitreolysis (PVL)
Number analyzed (Participants) | 35
Age, Continuous [Mean (Standard Deviation); unit: years] | 69 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 11
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 27
  Hispanic or Latino | 5
  non-Hispanic Black/African American | 3
Diabetes Type [Count of Participants; unit: Participants]
  No | 27
  Type 2 | 8
E-ETDRS visual acuity letter score [Mean (Standard Deviation); unit: units on a scale] — Measure Description: Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity.
  units on a scale | 55.8 (14)
Intraocular pressure [Mean (Standard Deviation); unit: mmHg] | 16 (3)
Lens Status on Clinical Exam [Number; unit: Eyes]
  Phakic (natural lens) | 28
  Prosthetic intraocular lens | 7
Epiretinal membrane in central subfield [Number; unit: Eyes] — Randomization stratification factor
  Eyes | 1
Width of vitreomacular attachment that extends within the central subfield [Median (Inter-Quartile Range); unit: Microns] | 325 [185 to 496]
Loss of ellipsoid zone integrity in central subfield [Number; unit: Eyes] | 35
Loss of ellipsoid zone integrity in foveal center [Number; unit: Eyes] | 35
Macular hole width at narrowest point [Median (Inter-Quartile Range); unit: micron] | 79 [39 to 111]

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Eyes With Macular Hole Closure of Inner Retinal Layers Without Rescue Vitrectomy
Time Frame: at 8 weeks
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis (PVL)
Number analyzed (Participants) | 35
Number analyzed (Eyes) | 35
Eyes | 10

2. Secondary Outcome: Mean Change in E-ETDRS Visual Acuity Letter Score From Baseline
Description: Best-corrected visual acuity following protocol-defined refraction. Visual Acuity was measured with the Electronic Early Treatment Diabetic Retinopathy Study (E-ETDRS) visual acuity test on a scale from 100 letters (Snellen equivalent of 20/10) to 0 letters (Snellen equivalent <20/800). Higher scores indicate better visual acuity and lower scores indicate worse visual acuity.
Time Frame: Baseline to 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis (PVL)
Number analyzed (Participants) | 35
Number analyzed (Eyes) | 35
units on a scale | -1.5 (25.6)

3. Secondary Outcome: E-ETDRS Visual Acuity Letter Score
Description: as for outcome 2
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis (PVL)
Number analyzed (Participants) | 35
Number analyzed (Eyes) | 35
units on a scale | 54.2 (23.8)

4. Secondary Outcome: Number of Eyes With Rescue Treatment Before the 8-week Visit
Time Frame: up to 8 Weeks
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis (PVL)
Number analyzed (Participants) | 35
Number analyzed (Eyes) | 35
Eyes | 12

5. Secondary Outcome: Macular Hole Closure Without Rescue Vitrectomy
Time Frame: 8 Weeks
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis (PVL)
Number analyzed (Participants) | 35
Number analyzed (Eyes) | 35
Eyes | 10

6. Secondary Outcome: Macular Hole Closure With Rescue Vitrectomy
Time Frame: 8 weeks
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis (PVL)
Number analyzed (Participants) | 35
Number analyzed (Eyes) | 35
Eyes | 10

7. Secondary Outcome: No Macular Hole Closure and no Rescue Vitrectomy
Time Frame: 8 weeks
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis (PVL)
Number analyzed (Participants) | 35
Number analyzed (Eyes) | 35
Eyes | 13

8. Secondary Outcome: No Macular Hole Closure Despite Rescue Vitrectomy
Time Frame: 8 weeks
Measure: Number; unit: Eyes
Units Other Than Participants: Eyes
Arm/Group | Pneumatic Vitreolysis (PVL)
Number analyzed (Participants) | 35
Number analyzed (Eyes) | 35
Eyes | 2

ADVERSE EVENTS:
Time Frame: 24-Weeks
Arm/Group | Pneumatic Vitreolysis (PVL)
All-Cause Mortality (participants affected / at risk) | 0/35
Serious Adverse Events (participants affected / at risk) | 5/35
Other Adverse Events (participants affected / at risk) | 15/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumatic Vitreolysis (PVL) (N=35)
Retinal tear (Eye disorders) | 3 (3)
Rhegmatogenous retinal detachment (Eye disorders) | 4 (4)
Embolism - blood clot (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pneumatic Vitreolysis (PVL) (N=35)
Anterior chamber cell (Eye disorders) | 1 (1)
Anterior chamber opacity (Eye disorders) | 1 (1)
Cataract (Eye disorders) | 1 (1)
Corneal abrasion (Eye disorders) | 1 (1)
Corneal defect (Eye disorders) | 1 (1)
Corneal edema (Eye disorders) | 1 (1)
Corneal pigmentation (Eye disorders) | 1 (1)
Dry eye (Eye disorders) | 1 (1)
Eye irritation (Eye disorders) | 1 (1)
Eye itching (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Floaters (Eye disorders) | 1 (1)
Macular hole (Eye disorders) | 2 (2)
Ocular discomfort (Eye disorders) | 1 (1)
Ocular hypertension (Eye disorders) | 4 (4)
Posterior capsule opacification (Eye disorders) | 1 (1)
Posterior vitreous detachment (Eye disorders) | 2 (2)
Red eye (Eye disorders) | 1 (1)
Subconjunctival hemorrhage (Eye disorders) | 3 (3)
Visual acuity decreased (Eye disorders) | 1 (1)
Visual flashes (Eye disorders) | 1 (1)
Vitreous debris (Eye disorders) | 1 (1)
Vitreous hemorrhage (Eye disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT03677869/Prot_000.pdf
  • Statistical Analysis Plan (2021-01-19): https://cdn.clinicaltrials.gov/large-docs/69/NCT03677869/SAP_001.pdf
  • Informed Consent Form (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT03677869/ICF_002.pdf